CLINICAL TRIAL: NCT01633294
Title: Antibiotic Prophylaxis in Prelabor Rupture of Membranes at Term - a Randomized Controlled Trial
Brief Title: Antibiotic Prophylaxis in Prelabor Rupture of Membranes at Term
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Hospital de Santa Maria, Portugal (Other)
Responsible Party: Principal Investigator, Filipa Faria Vaz Passos, Principal investigator, Hospital de Santa Maria, Portugal
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 335/08 - 28/07/08
Record Dates: First submitted 2012-06-23; First posted 2012-07-04 (Estimated); Last update posted 2016-11-28 (Estimated); Status verified 2016-11

CONDITIONS: Chorioamnionitis; Puerperal Endometritis; Neonatal Early Onset Sepsis; Neonatal Meningitis; Neonatal Pneumonia
Keywords: premature rupture of membranes; term pregnancy; chorioamnionitis; endometritis; neonatal sepsis; antibiotic prophylaxis
MeSH Terms: conditions — Chorioamnionitis; Neonatal Sepsis; Fetal Membranes, Premature Rupture; Endometritis | interventions — Ampicillin; Gentamicins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Antibiotic group (Active Comparator): women submitted to antibiotic prophylaxis
  Interventions: Drug: Ampicillin + gentamicin
- Control group (No Intervention)

INTERVENTIONS:
Drug: Ampicillin + gentamicin — ampicillin 1 g every six hours and gentamicin 240 mg every day intravenously
  Arms: Antibiotic group

SUMMARY:
The aims of this study are to determine whether antibiotics administered routinely in women presenting with premature rupture of membranes later than the 37+0 weeks of gestation can alter the rate of maternal and neonatal infection and to compare these rates between prompt (< 12 hour) and delayed (≥ 12 hour) induction in the group of patients not submitted to antibiotic prophylaxis.

ELIGIBILITY:
Inclusion Criteria:

* term (≥ 37+0 weeks) singleton pregnancy
* a vertex presentation
* ruptured membranes for less than 12 hours
* negative Group B Streptococcus (GBS) culture performed between 35 and 37 weeks

Exclusion Criteria:

* active labor
* absence of GBS culture or indication for GBS antibiotic prophylaxis (such as maternal GBS colonization between 35 and 37 weeks, GBS bacteriuria, prior infant with GBS sepsis)
* contraindication to expectant management (such as fetal distress, meconium staining of the amniotic fluid or chorioamnionitis) or to vaginal delivery

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 161 (Actual)
Dates: Start 2008-10; Primary Completion 2011-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
neonatal infection rate | participants will be followed for the duration of hospital stay, an expected average of 3 days
  neonatal infection rate includes early onset sepsis, meningitis and pneumonia
maternal infection rate | participants will be followed for the duration of hospital stay, an expected average of 3 days
  maternal infection rate includes chorioamnionitis or puerperal endometritis

SECONDARY OUTCOMES:
comparison of the infection rates between prompt and delayed induction | participants will be followed for the duration of hospital stay, an expected average of 3 days
  rate of maternal and neonatal infection between prompt (<12h) and delayed induction (≥12h) in the group of patients not submitted to antibiotic prophylaxis

CONTACTS AND LOCATIONS:
Overall Officials: Filipa Faria Vaz Passos, Dr, Principal Investigator — Santa Maria Hospital
Locations (1):
- Hospital Santa Maria, Lisbon, Portugal

REFERENCES:
- [Derived] Passos F, Cardoso K, Coelho AM, Graca A, Clode N, Mendes da Graca L. Antibiotic prophylaxis in premature rupture of membranes at term: a randomized controlled trial. Obstet Gynecol. 2012 Nov;120(5):1045-51. doi: 10.1097/aog.0b013e31826e46bc. PMID 23090521